CLINICAL TRIAL: NCT00597064
Title: Inflammatory, Functional and Image Composite Measure to Define Asthma Control
Acronym: APITA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ana Luisa Godoy Fernandes, Federal University of Sao Paulo- Respiratory Division
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APITA; FAPESP PROTOCOL; 2005/04714-1
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2007-11

CONDITIONS: Asthma
Keywords: asthma; asthma control questionnaire; oral corticosteroid; air trapping; AQLQ; control; quality of life
MeSH Terms: conditions — Asthma | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: prednisone — oral prednisone 40 mg/day for 15 +/- 5 days
  Other Names: prednisone or placebo radom assigned

SUMMARY:
The goals of control status of asthma have been changed with the improvement of its management as a chronic disease; many steps should be taken to achieve asthma control as defined by the GINA/NIH guidelines. There are good results with single variables, but overall asthma control should be addressed in different ways. Most traditional clinical studies provide an incomplete assessment of disease control, despite good clinical practice. The association of inhaled corticosteroid (IC) and long-action beta 2 agonist (LABA) has already showed their efficacy to reduce asthma symptoms, exacerbations and cost for moderate and severe asthma patients as well as the improvement in their quality of life. On the other hand, even with the use of first line maintenance medication, as recommended by guidelines, some asthmatic patients fail in obtaining a total control of the disease. This lack of efficacy, led us to hypothesize, that these patients who fail in response, would present chronic and fixed airway obstruction as a consequence of persistent inflammation and airway remodeling. This study has the purpose of looking for an adequate composite measure to provide an indicator of overall asthma status more accurately and meaningfully as reflect of treatment effectiveness and disease control. For this, we will test by a randomized control trial if an additional oral corticosteroid treatment could modify spirometric and plethysmography values, nasal and low airway cytology and HRCT (to evaluate small airway) in regularly treated stable asthma patients who have a positive bronchodilator response.

DETAILED DESCRIPTION:
To evaluate the achievement of asthma control status in asthmatic patients, regularly treated with IC + LABA to answer the following questions:

i. Is it possible to improve the pulmonary function (spirometry and plethysmography) of stable asthma patients, regularly treated with IC + LABA, who have a positive bronchodilator response, with the introduction of oral steroid?

ii. What is the relationship among nasal, induced sputum and blood cytology, as a tool to observe inflammatory airway expression, in controlled and total controlled asthma patients? What will be these values response if oral steroids have been introduced?

iii. What is the correlation between pulmonary volumes and airways inflammation to evaluate severity and control status in asthmatic patients, using plethysmography and HRCT? What will be these values response if oral steroids have been introduced?

ELIGIBILITY:
Inclusion criteria:

* A documented clinical asthma history at least for a period of six months
* Regular treatment (IC + LABA) at least for a period of three months
* Controlled symptoms score defined by GINA 2002 criteria (daytime symptoms < 2 days a week and no night time symptoms in the last 15 days) or complete absence of chronic symptoms
* None or minimal exacerbations without emergency visits
* Absent or a minimal usage bronchodilator rescue, side effects of medication and limitation to exercises
* Documented airway reversibility of 200 ml and 7% based on predicted values of VEF1

Exclusion Criteria:

* Having a smoking history of 5 pack/years or more; having other known chronic pulmonary diseases; having side effect to oral corticosteroid
* Having an upper or lower respiratory tract infection within 4 weeks of visit 0
* Unable to do the tests involved in the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Asthma control status characterized by nocturnal and diurnal symptom score FEV1,total lung capacity in plethysmography and reducing the air-tapping in HRCT. | 30 days

SECONDARY OUTCOMES:
Quality of life, Sputum and nasal cytology, adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ana Luisa G Fernandes, MD, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Rua Botucatu 740 3 ° and - Pneumologia, São Paulo, São Paulo, Brazil